CLINICAL TRIAL: NCT07380646
Title: A Single-Arm, Phase II, Multicenter Clinical Trial to Evaluate the Efficacy of Leucogen in Preventing the Risk of Ribociclib-Associated Neutropenia in Patients With Hormone Receptor-Positive, HER2-Negative Early Breast Cancer
Brief Title: the Efficacy of Leucogen in Preventing the Risk of Ribociclib-Associated Neutropenia in Early Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-1460
Record Dates: First submitted 2025-12-22; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Leucogen; Ribociclib; Neutropenia (Low White Blood Cell Count); Breast Cancer
MeSH Terms: conditions — Neutropenia; Leukopenia; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-Arm, Phase II, Multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leucogen combined with Ribociclib (Kisqali®) and Endocrine Therapy (e.g., Letrozole, Anastrozol) (Experimental): The experimental arm receives ribociclib at the standard dose (orally, 400mg, once daily on days 1-21 of a 28-day cycle) combined with a specified endocrine therapy (e.g., letrozole or anastrozole) plus leucogen (40mg orally three times daily on days 8-28 of a 28-day cycle).
  Interventions: Drug: Treat Regimen

INTERVENTIONS:
Drug: Treat Regimen — leucogen combined with ribociclib and endocrine therapy

SUMMARY:
This study is a multicenter, single-arm, open-label Phase II exploratory clinical trial designed to evaluate whether prophylactic use of leucogen can reduce the incidence of Grade 3 or higher neutropenia in early-stage HR+/HER2- breast cancer patients receiving ribociclib combined with endocrine therapy. The study plans to enroll 97 patients using a Simon two-stage design, with the primary endpoint being the incidence of severe neutropenia within 4 treatment cycles (4 months) after initiation. Secondary endpoints include the incidence of all-grade neutropenia, febrile neutropenia, ribociclib treatment intensity, and safety. The study will systematically assess the preventive efficacy and safety of leucogen to provide a basis for subsequent Phase III randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed and dated the informed consent form.
2. Age > 18 years at the time of signing informed consent.
3. The patient is a female with known menopausal status at the time of signing informed consent or initiation of adjuvant endocrine therapy (whichever is earlier). Postmenopausal status is defined as: bilateral oophorectomy, age > 60 years, or age < 60 years with amenorrhea ≥ 12 months (in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression), and follicle-stimulating hormone and plasma estradiol levels within the local postmenopausal normal range.
4. Histologically confirmed unilateral primary invasive breast cancer, with the date of initial cytological or histological diagnosis within 18 months before enrollment. Patients with multicentric and/or multifocal tumors are eligible if all pathologically examined lesions meet criteria 5 and 6 below.
5. Estrogen receptor (ER) and/or progesterone receptor (PgR) positivity in the breast cancer, based on the most recent analyzed tissue sample from the local laboratory.
6. HER2-negative breast cancer, defined as negative by in situ hybridization or immunohistochemistry (IHC) status of 0 or 1+. If IHC is 2+, a negative in situ hybridization result is required to confirm HER2-negative status (based on the most recent analyzed tissue sample from the local laboratory).
7. The patient has undergone surgical resection with complete tumor removal, negative microscopic margins on the final surgical specimen, and belongs to one of the following categories:

   Anatomic Stage II, with any of the following: T0-2N1, T3N0, T2N0 with Grade 2 and Ki-67 ≥ 20%, T2N0 with Grade 2 and high-risk genomic assay result, T2N0 with Grade 3.

   Anatomic Stage III. High-risk genomic assay is defined as Oncotype DX Recurrence Score ≥ 26, or high-risk group by Prosigna PAM50, MammaPrint, or EndoPredict.
8. If clinically indicated, the patient has completed adjuvant and/or neoadjuvant chemotherapy according to guidelines before screening.
9. If clinically indicated, the patient has completed adjuvant radiotherapy according to guidelines before screening.
10. The patient has no contraindications to the adjuvant endocrine therapy in the trial and plans to receive endocrine therapy for 5 years or longer starting from the randomization date.
11. The patient may have received any standard neoadjuvant endocrine therapy at the time of signing informed consent, but enrollment must occur within 12 months of the first endocrine therapy initiation. Note: Endocrine therapy for ovarian suppression or short-term fertility preservation is not considered neoadjuvant/adjuvant endocrine therapy. If the patient is using tamoxifen as adjuvant endocrine therapy, a washout period of 5 half-lives is required before enrollment, during which the patient may take an aromatase inhibitor.
12. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
13. Adequate bone marrow and organ function defined by meeting the following local laboratory values:

    Absolute neutrophil count ≥ 1.5 × 10⁹/L Platelet count ≥ 100 × 10⁹/L Hemoglobin ≥ 9.0 g/dL Estimated glomerular filtration rate (eGFR) by MDRD formula ≥ 30 mL/min/1.73m² Alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN) Aspartate aminotransferase (AST) ≤ 2.5 × ULN Serum total bilirubin < ULN; or for patients with documented Gilbert's syndrome: total bilirubin ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN International normalized ratio (INR) ≤ 1.5 (unless the patient is on anticoagulant therapy and the INR is within the expected therapeutic range for that anticoagulant within 7 days before enrollment)
14. The following laboratory parameters must be within normal limits or corrected to normal range with supplementation (corrected local laboratory values should be recorded as normal):

    Sodium Potassium Magnesium Total calcium (corrected for serum albumin)
15. Standard 12-lead electrocardiogram assessed by the local institution meeting the following:

    Screening QTcF interval < 450 ms Resting heart rate 50-90 beats per minute (determined by ECG)
16. The patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.
17. Females of childbearing potential must have a negative serum pregnancy test (for β-hCG) within 14 days before enrollment. Females of childbearing potential must be willing to use highly effective contraception. A female is considered to be of childbearing potential unless she has had natural amenorrhea for 12 months with appropriate clinical features (i.e., age-appropriate history of vasomotor symptoms), or has undergone bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before randomization. In the case of oophorectomy alone, only after the female's reproductive status has been confirmed by subsequent hormone level assessment is she considered not of childbearing potential.
18. Contraception must be continued during the trial treatment and for 21 days after treatment discontinuation.

Exclusion Criteria:

1. Previous treatment with any CDK4/6 inhibitor.
2. Use of tamoxifen, raloxifene, or aromatase inhibitors for breast cancer risk reduction ("chemoprevention") and/or osteoporosis treatment within 2 years before signing informed consent.
3. Prior anthracycline cumulative dose reaching or exceeding: doxorubicin 450 mg/m², or epirubicin 900 mg/m².
4. Known hypersensitivity to any excipient of ribociclib and/or the endocrine therapy and/or leucogen (e.g., rare hereditary galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, or soy allergy).
5. Evidence of distant metastasis of breast cancer beyond regional lymph nodes (AJCC 8th edition Stage IV) and/or recurrence after curative surgery.
6. Concurrent use of other anticancer therapies, except adjuvant endocrine therapy.
7. Major surgery, chemotherapy, or radiotherapy within 14 days before enrollment.
8. Clinical and laboratory acute toxicities related to prior anticancer therapy have not recovered to Grade 1 or lower (per NCI CTCAE version 4.03) on the day of enrollment. Exceptions: alopecia and amenorrhea of any grade are allowed.
9. Current invasive malignancy, or previous invasive malignancy completed treatment within 2 years before signing informed consent. Note: Patients with past or concurrent in situ malignancy are eligible if they have undergone adequate curative treatment before enrollment.
10. Known history of human immunodeficiency virus (HIV) infection.
11. Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
12. Clinically significant, uncontrolled cardiac disease and/or cardiac repolarization abnormalities, including any of the following:

    Documented history of myocardial infarction, angina, symptomatic pericarditis, or coronary artery bypass grafting within 6 months before trial enrollment.

    Documented cardiomyopathy. Left ventricular ejection fraction < 50% as measured by multigated acquisition scan or echocardiography.

    Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or presence of any of the following risk factors: risk factors for torsades de pointes including uncorrected hypokalemia or hypomagnesemia, history of heart failure, or history of clinically significant/symptomatic bradycardia. Concurrent use of medications known to prolong the QT interval and/or known to cause TdP that cannot be discontinued or switched to a safe alternative (e.g., within 5 half-lives or 7 days before starting trial treatment). Inability to determine QTcF interval.

    Clinically significant arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular block (e.g., bifascicular block, Mobitz type II, and third-degree AV block).

    Uncontrolled hypertension with systolic blood pressure > 160 mmHg.
13. Use of any of the following within 7 days before enrollment:

    Concomitant medications, herbal supplements, and/or fruits (e.g., grapefruit, pomelo, carambola, Seville oranges) and their juices that are known potent inhibitors or inducers of CYP3A4/5.

    Drugs with a narrow therapeutic window that are predominantly metabolized by CYP3A4/5.
14. Systemic corticosteroid therapy within ≤ 2 weeks before starting trial treatment, or not fully recovered from side effects of such therapy.
15. Treatment with immunomodulators or other drugs affecting leukocytes (e.g., thymosin, batyl alcohol, IL-11, GM-CSF, G-CSF) within ≤ 4 weeks before starting trial treatment.
16. Impaired gastrointestinal function or gastrointestinal disease that may significantly alter absorption of oral trial drugs (e.g., uncontrolled ulcerative disease, uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, or small bowel resection).
17. Any other concurrent severe and/or uncontrolled medical condition that, in the investigator's judgment, would pose an unacceptable safety risk, contraindicate participation in the clinical trial, or affect compliance with the protocol (e.g., chronic pancreatitis, chronic active hepatitis, cirrhosis or any other significant liver disease, active untreated or uncontrolled fungal, bacterial or viral infection, active infection requiring systemic antimicrobial therapy, etc.), or would limit life expectancy to ≤ 5 years.
18. Participation in another interventional study with investigational product treatment (or use of an investigational device) within 30 days before enrollment, or within 5 half-lives of the investigational product (whichever is longer).
19. Complete blood count within 1 week before ribociclib administration showing white blood cell or neutrophil count below the lower limit of normal of the testing institution.
20. Pregnancy or lactation, or planning to become pregnant or breastfeed during the trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
incidence of severe neutropenia | From enrollment to the end of treatment at 16 weeks
  Complete blood count (CBC) should be performed on Day 1 and Day 21 of each treatment cycle. A decrease in the absolute neutrophil count (ANC) to < 1000-500/mm³ (which is equivalent to < 1.0-0.5 × 10⁹/L) is defined as severe neutropenia.

IPD SHARING:
Plan to Share IPD: No